CLINICAL TRIAL: NCT07198360
Title: Incidence, Risk Factors, and Outcomes of Intraventricular Hemorrhage in Preterm Infants Admitted to the NICU
Brief Title: Outcome of Intraventricular Hemorrhage in Preterm Infants
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Romany Nady Isaac Ayad, Pediatric resident, Assiut University
Other Study IDs: IVH in preterm infants
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Intraventricular Hemorrhage of Prematurity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — Not found

SUMMARY:
To determine the incidence and grading of IVH among preterm neonates in the NICU.

* To identify maternal and neonatal risk factors associated with IVH.
* To assess short-term outcomes (mortality, Hydrocephalus, need for neurosurgical intervention, seizures, length of Hospital stay).

DETAILED DESCRIPTION:
Intraventricular hemorrhage (IVH) is described as bleeding that occurs within and surrounding the brain ventricles, which contain cerebrospinal fluid . IVH is one of the most severe complications affecting preterm newborns globally, frequently leading to poor prognoses and potential mortality due to both short- and long-term neurodevelopmental consequences. The risk is markedly elevated for preterm newborns with a short gestational age, as roughly 15-20% of those born prior to 32 weeks of gestation are at the greatest risk of suffering a severe form of intraventricular hemorrhage . In term newborns, IVH occurs with an incidence of 5.5%, primarily due to perinatal head trauma, birth hypoxia, or coagulation disorders .

The IVH is diagnosed using cranial ultrasound (CUS), which is performed within the first 72 hours of life and repeated as clinically indicated. The IVH grade will be classified according to the Papile classification, which includes Grades I, II, III, and IV . Grades I and II were classified as mild intraventricular hemorrhage (IVH), whereas grades III and IV were classified as severe IVH. Grade IV IVH is now designated as periventricular hemorrhage infarction or parenchymal hemorrhage in recent years .

The risk factors for IVH include acute placental inflammation, elevated leukocyte count within the first 72 hours post-birth, increased white blood cell levels, and male sex. Additional risk factors for IVH encompass prematurity, low birthweight (LBW), prolonged mechanical ventilation, a low 5-minute Apgar score, hypoxia-related injury, hypothermic ischemia, pneumothorax, thrombocytopenia, antenatal maternal hemorrhage, maternal infection or inflammation, sepsis, hypotension, hypoxia, hypercapnia, seizures, patent ductus arteriosus (PDA), infection, respiratory distress, and genetic predispositions .

IVH in neonates, particularly preterm infants, often presents with nonspecific clinical signs such as apnea, bradycardia, hypotonia, bulging fontanelle, seizures, or a sudden drop in hematocrit. Some cases may be clinically silent, making routine screening essential . The diagnosis is primarily made using transcranial ultrasound (cranial sonography), which is a non-invasive, bedside imaging tool capable of detecting IVH grades, ventricular dilation, and parenchymal involvement through the anterior fontanelle. Outcomes vary depending on the severity (graded IIV), with lower grades (III) often resolving without long-term consequences, while higher grades (IIIIV) are associated with complications such as post-hemorrhagic hydrocephalus, cerebral palsy, developmental delay, and increased mortality. Early detection through serial ultrasound monitoring plays a critical role in management and prognosis .

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates < 34 weeks of gestation
* Birth weight < 1500g
* Admitted to NICU within 24 hours of birth

Exclusion Criteria:

* Major congenital malformations (especially CNS anomalies)
* Severe perinatal asphyxia
* Neonates with congenital infections (TORCH)

Max Age: 28 Days | Sex: All
Age Groups: Child
Study Population: All with the required Criteria
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
. To determine the incidence of IVH in preterm infants within the first 7 days of life using cranial ultrasound. . To assess the grade of IVH (Papile classification I-IV) in preterm infants based on cranial US findings. | Baseline
  Outcome of intraventricular haemorrhage in preterm infants

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parodi A, Govaert P, Horsch S, Bravo MC, Ramenghi LA; eurUS.brain group. Cranial ultrasound findings in preterm germinal matrix haemorrhage, sequelae and outcome. Pediatr Res. 2020 Mar;87(Suppl 1):13-24. doi: 10.1038/s41390-020-0780-2. PMID 32218535
- [Background] Kolnik SE, Upadhyay K, Wood TR, Juul SE, Valentine GC. Reducing Severe Intraventricular Hemorrhage in Preterm Infants With Improved Care Bundle Adherence. Pediatrics. 2023 Sep 1;152(3):e2021056104. doi: 10.1542/peds.2021-056104. PMID 37609772
- [Background] Legge N, Lutz T, Wocadlo C, Rieger I. Long-term neurodevelopmental outcome in preterm infants with intraventricular haemorrhage. J Paediatr Child Health. 2022 Oct;58(10):1797-1802. doi: 10.1111/jpc.16108. Epub 2022 Jul 15. PMID 35837759